CLINICAL TRIAL: NCT04305054
Title: A Phase 1/2 Open-Label Rolling-Arm Umbrella Platform Design of Investigational Agents With or Without Pembrolizumab or Pembrolizumab Alone in Participants With Melanoma (KEYMAKER-U02): Substudy 02B
Brief Title: Substudy 02B: Safety and Efficacy of Pembrolizumab in Combination With Investigational Agents or Pembrolizumab Alone in Participants With First Line (1L) Advanced Melanoma (MK-3475-02B/KEYMAKER-U02)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-02B; MK-3475-02B (Other: MSD); KEYMAKER-U02 (Other: MSD); 2023-506313-21-00 (Registry Identifier: EU CT); U1111-1293-5644 (Registry Identifier: UTN); 2019-003977-24 (EudraCT Number)
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Melanoma
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death ligand 1 (PD-L1, PDL1); T cell immunoreceptor with immunoglobulin and immunoreceptor tyrosine receptor motif domains (TIGIT); Cytotoxic T lymphocyte associated protein 4 (CTLA4)
MeSH Terms: conditions — Melanoma; Parkinson Disease 4, Autosomal Dominant Lewy Body; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- Pembrolizumab + Vibostolimab (Experimental): Participants will receive pembrolizumab intravenously (IV) plus vibostolimab IV at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: Vibostolimab
- Pembrolizumab (Active Comparator): Participants will receive pembrolizumab IV at a specified dose on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab
- Coformulation Pembrolizumab/Quavonlimab (Experimental): Participants will receive coformulation of pembrolizumab and quavonlimab (MK-1308A) IV at a specified dose on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: Pembrolizumab/Quavonlimab
- Coformulation Pembrolizumab/Quavonlimab + Lenvatinib (Experimental): Participants will receive coformulation of pembrolizumab and quavonlimab IV plus lenvatinib orally at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Pembrolizumab; Biological: Pembrolizumab/Quavonlimab; Drug: Lenvatinib
- Coformulation Favezelimab/Pembrolizumab (Experimental): Participants will receive cofomulation of favezelimab + pembrolizumab (MK-4280A) IV at specified dose on specified days every 3 weeks (Q3W) for up to approximately 2 years
  Interventions: Biological: Favezelimab/Pembrolizumab
- Coformulation Favezelimab/Pembrolizumab + All-trans Retinoic Acid (ATRA) (Experimental): Participants will receive coformulation of favezelimab and pembrolizumab IV Q3W for up to 35 cycles, plus ATRA orally (for 3 days surrounding each infusion of MK-4280A, including Days 1, 2, and 3 of Cycle 1 and on Days -1, 1, and 2 of all subsequent cycles).
  Interventions: Drug: ATRA
- Coformulation Favezelimab/Pembrolizumab + Vibostolimab (Experimental): Participants will receive coformulation of favezelimab and pembrolizumab (MK-4280A) IV and vibostolimab IV at specified doses on specified days for a total treatment duration of up to approximately 2 years.
  Interventions: Biological: Vibostolimab; Biological: Favezelimab/Pembrolizumab

INTERVENTIONS:
Biological: Pembrolizumab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-3475; KEYTRUDA®
  Arms: Coformulation Pembrolizumab/Quavonlimab; Coformulation Pembrolizumab/Quavonlimab + Lenvatinib; Pembrolizumab; Pembrolizumab + Vibostolimab
Biological: Vibostolimab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-7684
  Arms: Coformulation Favezelimab/Pembrolizumab + Vibostolimab; Pembrolizumab + Vibostolimab
Biological: Pembrolizumab/Quavonlimab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-1308A
  Arms: Coformulation Pembrolizumab/Quavonlimab; Coformulation Pembrolizumab/Quavonlimab + Lenvatinib
Drug: Lenvatinib — Administered via oral capsule at a specified dose on specified days
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Coformulation Pembrolizumab/Quavonlimab + Lenvatinib
Biological: Favezelimab/Pembrolizumab — Administered via IV infusion at a specified dose on specified days
  Other Names: MK-4280A
  Arms: Coformulation Favezelimab/Pembrolizumab; Coformulation Favezelimab/Pembrolizumab + Vibostolimab
Drug: ATRA — Administered via oral capsule at a specified dose on specified days
  Arms: Coformulation Favezelimab/Pembrolizumab + All-trans Retinoic Acid (ATRA)

SUMMARY:
Substudy 02B is part of a larger research study where researchers are looking for new ways to treat advanced melanoma that has not been treated before. The larger study is the umbrella study. Researchers want to know if adding other treatments to pembrolizumab can treat advanced melanoma. The goals of this study are to learn:

* About the safety and how well people tolerate pembrolizumab given with other treatments
* How many people have melanoma that responds (gets smaller or goes away) to treatment

DETAILED DESCRIPTION:
With Amendment 6, all arms are closed to enrollment. Participants in arms 2 (pembrolizumab), 3 (coformulation pembrolizumab/quavonlimab), and 4 (coformulation pembrolizumab/quavonlimab + lenvatinib) who complete study treatment or otherwise meet end of treatment (EOT) criteria will be discontinued from the study after completing the EOT visit and any required safety follow-up visits. Participants in arm 6 (coformulation favezelimab/pembrolizumab + All-trans Retinoic Acid [ATRA]) will discontinue ATRA and participants in arms 5 and 6 can continue on coformulation favezelimab/pembrolizumab or pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Has histologically or cytologically confirmed melanoma
* Has unresectable Stage III or Stage IV melanoma, not amenable to local therapy
* Has been untreated for advanced disease.
* Has provided a tumor biopsy
* If capable of producing sperm, male participants agree to the following during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention (7 days):

  * Abstains from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) and agrees to remain abstinent OR
  * Uses contraception unless confirmed to be azoospermic
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a WOCBP OR
  * Is a WOCBP and Uses a contraceptive method that is highly effective, with low user dependency, or be abstinent from penile-vaginal intercourse as their preferred and usual lifestyle (abstinent on a long-term and persistent basis) during the intervention period and for at least the time needed to eliminate each study intervention after the last dose of study intervention. The length of time required to continue contraception for each study intervention is:
  * MK-4280A: 120 days
  * MK-1308A: 120 days
  * MK-7684: 50 days
  * MK-3475: 120 days
  * Lenvatinib: 30 days
  * ATRA: 30 days
* Has adequate organ function
* Has resolution of toxic effect(s) of the most recent prior therapy to Grade 1 or less (except alopecia and Grade 2 neuropathy)

Exclusion Criteria:

* Has a diagnosis of immunodeficiency or is receiving immunosuppressive therapy within 7 days before the first dose of study intervention
* Has a known additional malignancy that is progressing or requires active treatment within the past 2 years
* Has known central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has ocular or mucosal melanoma
* Has an active autoimmune disease that has required systemic treatment in the past 2 years
* Has an active infection requiring systemic therapy
* Has known history of human immunodeficiency virus (HIV)
* Has history of Hepatitis B or known Hepatitis C virus infection
* Has a history of (noninfectious) pneumonitis
* Has a history of active tuberculosis (TB)
* Has received prior systemic anticancer therapy within 4 weeks prior to randomization
* Has received prior radiotherapy within 2 weeks of first dose of study intervention
* Has had major surgery <3 weeks prior to first dose of study intervention
* Has received a live vaccine within 30 days before the first dose of study intervention
* Has participated in a study of an investigational agent within 4 weeks prior to the first dose of study intervention
* Has had an allogeneic tissue/solid organ transplant
* Has a known psychiatric or substance abuse disorder that would interfere with requirements of the study
* Participants who receive lenvatinib have the following additional exclusion criteria:

  * Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula
  * Has radiographic evidence of encasement of invasion of a major blood vessel, or of intratumoral cavitation
  * Has clinically significant hemoptysis or tumor bleeding within 2 weeks prior to the first dose of study intervention
  * Has clinically significant cardiovascular disease within 12 months from first dose of study intervention
  * Has urine protein ≥1 g/24-hour.
  * Has presence of gastrointestinal condition including malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of lenvatinib

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2026-04-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who experience a dose-limiting toxicity (DLT): Safety lead-in phase | Up to ~3 weeks
  The percentage of participants who experience 1 or more protocol-defined DLTs during the safety lead-in period will be reported.
Percentage of participants who experience an adverse event (AE): Safety lead-in | Up to ~3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience an AE during the safety lead-in period will be reported.
Percentage of participants who discontinue study treatment due to an AE: Safety lead-in | Up to ~3 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study treatment due to an AE during the safety lead-in will be reported.
Percentage of participants who experience an adverse event (AE) | Up to ~28 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who experience an AE will be reported.
Percentage of participants who discontinue study treatment due to an AE | Up to ~24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants who discontinue study treatment due to an AE will be reported.
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors 1.1 (RECIST 1.1) | Up to ~30 months
  ORR is defined as the percentage of participants in the analysis population who have a complete response (CR: disappearance of all target lesions) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters). Responses are according to RECIST 1.1 as assessed by blinded independent central review (BICR). RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

SECONDARY OUTCOMES:
Duration of Response (DOR) per RECIST 1.1 | Up to ~30 months
  For participants in the analysis population who demonstrate a confirmed CR (disappearance of all target lesions) or confirmed PR (at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum of diameters), DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death due to any cause, whichever occurs first. Responses are according to RECIST 1.1 as assessed by BICR. RECIST 1.1 has been modified for this study to include a maximum of 10 target lesions and a maximum of 5 target lesions per organ.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (60):
- United States (15):
  - The Angeles Clinic and Research Institute ( Site 2009), Los Angeles, California
  - UCLA Hematology & Oncology ( Site 2004), Los Angeles, California
  - Providence Saint John's Health Center ( Site 2010), Santa Monica, California
  - University of Colorado, Anschutz Cancer Pavilion ( Site 2012), Aurora, Colorado
  - University of Florida College of Medicine-UF Health Cancer Center/Clinical Trials Office ( Site 2026), Gainesville, Florida
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins ( Site 2022), Baltimore, Maryland
  - R.J. Zuckerberg Cancer Center ( Site 2032), Lake Success, New York
  - NYU Clinical Cancer Center ( Site 2002), New York, New York
  - Duke Cancer Institute ( Site 2005), Durham, North Carolina
  - Martha Morehouse Tower ( Site 2020), Columbus, Ohio
  - Oregon Health & Science University ( Site 2013), Portland, Oregon
  - University of Pennsylvania Abramson Cancer Center ( Site 2008), Philadelphia, Pennsylvania
  - West Cancer Center - East Campus ( Site 2014), Germantown, Tennessee
  - Mays Cancer Center ( Site 2025), San Antonio, Texas
  - Inova Schar Cancer Institute ( Site 2011), Fairfax, Virginia
- Argentina (3):
  - Clinica Adventista Belgrano-Oncology ( Site 2242), Caba., Buenos Aires
  - Instituto Alexander Fleming-Alexander Fleming ( Site 2243), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Finochietto ( Site 2245), Buenos Aires
- Australia (4):
  - Calvary Mater Newcastle-Medical Oncology ( Site 2404), Waratah, New South Wales
  - Melanoma Institute Australia ( Site 2402), Wollstonecraft, New South Wales
  - Tasman Oncology Research Pty Ltd ( Site 2403), Southport, Queensland
  - Fiona Stanley Hospital ( Site 2401), Murdoch, Western Australia
- Chile (5):
  - IC La Serena Research ( Site 2254), La Serena, Coquimbo Region
  - FALP-UIDO ( Site 2251), Santiago, Region M. de Santiago
  - Oncovida ( Site 2257), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 2252), Santiago, Region M. de Santiago
  - CIDO SpA-Oncology ( Site 2256), Temuco, Región de la Araucanía
- Colombia (2):
  - Clinica Colsanitas S.A, Sede Clínica Universitaria Colombia-Center Investigator ( Site 2261), Bogotá, Bogota D.C.
  - Fundación Valle del Lili ( Site 2265), Cali, Valle del Cauca Department
- France (6):
  - Hopital La Timone ( Site 2103), Marseille, Bouches-du-Rhone
  - CHU de Bordeaux- Hopital Saint Andre ( Site 2108), Bordeaux, Gironde
  - Institut Claudius Regaud ( Site 2105), Toulouse, Haute-Garonne
  - C.H. Lyon Sud ( Site 2102), Pierre-Bénite, Rhone
  - A.P.H. Paris, Hopital Saint Louis ( Site 2107), Paris
  - Gustave Roussy ( Site 2101), Villejuif, Île-de-France Region
- Greece (2):
  - General Hospital of Athens "Laiko"-First Department of Internal Medicine ( Site 2212), Athens, Attica
  - European Interbalkan Medical Center-Oncology Department ( Site 2211), Thessaloniki
- Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ ( Site 2221), Szeged, Csongrád megye, Hungary
- Israel (5):
  - HaEmek Medical Center ( Site 2703), Afula
  - Rambam Health Care Campus-Oncology ( Site 2704), Haifa
  - Hadassah Ein Karem Jerusalem ( Site 2702), Jerusalem
  - Rabin Medical Center-Oncology ( Site 2705), Petah Tikva
  - Chaim Sheba Medical Center ( Site 2701), Ramat Gan
- Italy (5):
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 2399), Milan
  - Istituto Europeo di Oncologia ( Site 2301), Milan
  - Istituto Nazionale Tumori Fondazione Pascale ( Site 2302), Napoli
  - Istituto Oncologico Veneto IRCCS ( Site 2355), Padua
  - Policlinico Le Scotte - A.O. Senese ( Site 2377), Siena
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 2233), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Early Clinical Trials Unit ( Site 2231), Gdansk, Pomeranian Voivodeship
- South Africa (5):
  - CANCERCARE LANGENHOVEN DRIVE ONCOLOGY CENTRE ( Site 2865), Port Elizabeth, Eastern Cape
  - Steve Biko Academic Hospital-Medical Oncology ( Site 2862), Pretoria, Gauteng
  - LIFE GROENKLOOF-Mary Potter Cancer Centre ( Site 2861), Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd-Research ( Site 2863), Sandton, Gauteng
  - Cape Town Oncology Trials ( Site 2864), Cape Town, Western Cape
- Spain (2):
  - HOSPITAL CLÍNIC DE BARCELONA-ICHMO- Clinic Institut of Haematological and Oncological diseases ( Site 2801), Barcelona, Catalonia
  - Hospital Universitario Ramón y Cajal ( Site 2802), Madrid, Madrid, Comunidad de
- Switzerland (3):
  - Hôpitaux Universitaires de Genève (HUG)-Oncology ( Site 2603), Geneva, Canton of Geneva
  - CHUV Centre Hospitalier Universitaire Vaudois ( Site 2602), Lausanne, Canton of Vaud
  - Universitaetsspital Zuerich ( Site 2601), Zuerich Flughafen, Canton of Zurich

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26251&tenant=MT_MSD_9011